CLINICAL TRIAL: NCT01294865
Title: The Plasma Levels of suPAR in Late-onset Neonatal Sepsis
Brief Title: Soluble Urokinase Plasminogen Activator Receptor (suPAR) in Late-onset Neonatal Sepsis
Acronym: suPAR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ankara University (Other)
Responsible Party: Saadet Arsan, Ankara University
Other Study IDs: Ankara University-02; Ankara University (Other Grant/Funding Number: Ankara University Research Fund (10B3330012))
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Last update posted 2011-02-14 (Estimated); Status verified 2009-12

CONDITIONS: Neonatal Sepsis
Keywords: Sepsis; late-onset; suPAR
MeSH Terms: conditions — Neonatal Sepsis; Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- septic: Infants having clinical suspected late-onset neonatal sepsis enrolled in the study. Blood samples for suPAR were obtained before initiating antibiotic treatment and at the end of the treatment with other laboratory tests.
- non-septic: Infants without any clinical or hematological septic signs. Blood samples will be taken only once.

SUMMARY:
The purpose of the study is to investigate the plasma levels of Soluble Urokinase Plasminogen Activator Receptor (suPAR) at the diagnosis and after treatment of sepsis, and to determine whether it has a diagnostic and prognostic value in late-onset neonatal sepsis.

DETAILED DESCRIPTION:
Infection is a leading cause of neonatal morbidity and mortality worldwide. The clinical presentation of neonatal infection is subtle and nonspecific. Microbiologic cultures of clinical specimens, the gold standard for diagnosis, have low sensitivity and are not available in time to influence initial therapy. Therefore, reliable and rapid in vitro tests are needed for early diagnosis and management of infection in neonates. suPAR, secreted from the cells (neutrophils, lymphocytes, macrophages, endothelial cells) has recently been reported to be a potential biomarker for several infection diseases. The levels of suPAR have not been studied in newborn infants yet.

ELIGIBILITY:
Inclusion Criteria:

* Infants with late-onset neonatal sepsis

Exclusion Criteria:

* Infants without parents' consent

Ages: 4 Days to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants in Ankara University neonatal intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Levels of suPAR in late-onset neonatal sepsis | three weeks
  Levels of suPAR will be dosed with suspicion of late-onset sepsis diagnosis at day 0 and at the end of the treatment. The evolution and the best cut-off values will be calculated for the diagnosis. Indices of sensibility, specificity, positive predictive value and negative predictive value will be calculated.

SECONDARY OUTCOMES:
Level of plasma C-reactive protein | three weeks
  Plasma C-reactive protein levels to confirm the diagnostic usefulness of suPAR measurements at diagnosis and end of the treatment
the white blood cell count | three weeks
  the white blood cell counts to confirm the diagnostic usefulness of suPAR measurements at diagnosis and end of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Saadet Arsan, Professor, Study Director — Ankara University
Locations (1):
- Ankara University Faculty of Medicine, Department of Pediatrics, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Okulu E, Arsan S, Akin IM, Ates C, Alan S, Kilic A, Atasay B. Serum Levels of Soluble Urokinase Plasminogen Activator Receptor in Infants with Late-onset Sepsis. J Clin Lab Anal. 2015 Sep;29(5):347-52. doi: 10.1002/jcla.21777. Epub 2014 Jul 10. PMID 25043869